CLINICAL TRIAL: NCT05139589
Title: The ENDOCARDITIS AUMC Data Collection : a Matched Cohort Study on Perioperative Coagulation in Conservatively and Surgically Treated Patients With Valvular Dysfunction, With and Without Infective Endocarditis
Brief Title: The ENDOCARDITIS AUMC Data Collection
Acronym: ENDO_AUMC
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jennifer Breel, Research Coordinator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_466#21.518
Record Dates: First submitted 2021-11-30; First posted 2021-12-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Endocarditis; Coagulation Disorder; Valve Disease, Heart
MeSH Terms: conditions — Endocarditis; Hemostatic Disorders; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infective endocarditis, surgical arm: Patients with infective endocardits requiring valve surgery
  Interventions: Other: None, observational
- Infective endocarditis, conservative arm: Patients with infective endocardits, not requiring valve surgery
  Interventions: Other: None, observational
- Valve disease, heart, surgically repaired: Patients requiring valve surgery
  Interventions: Other: None, observational

INTERVENTIONS:
Other: None, observational — Patients with infective endocarditis who do and do not undergo valve surgery compared with patientswithout endocarditis, who are operated on with similar valve surgery

SUMMARY:
The investigators will compare patients with and without infective ndocarditis undergoing valve surgery and evaluate factors that may help optimise perioperative care of these high-risk patients.

DETAILED DESCRIPTION:
The aim of this study is to examine the differences between patients with and without endocarditis who undergo cardiothoracic (valve) surgery. In addition, the investigators will look at the differences between endocarditis patients who undergo surgery, and those who are treated conservatively. The investigators will look at incidence and degree of perioperative coagulation abnormalities, as well as transfusion and coagulation factor requirements, heparin resistance, bleeding scores, predictive endocarditis mortality scores, vasopressor-inotrope scores, and relate these where possible to the pathogen causing IE. The investigators will also look at perioperative complications, in particular, thromboembolic events and mortality at 30 and 90 days, and at 1 year.

These outcomes may help optimise perioperative care for high-risk endocarditis patients, and in particular those undergoing valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Dutch or English speaking
* All patients with infective endocarditis admitted to Amsterdam UMC in the study period
* All patients with infective endocarditis scheduled for cardiac valve surgery compared to a matched cohort of patients scheduled for similar surgery due to non-infectious indication in Amsterdam UMC in the same period

Exclusion Criteria:

* Previous history of coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of two groups (a study group and a control group) of male and female patients, 18 years and older. The study group consists of all patients with infective endocarditis admitted to the Amsterdam UMC, in either location. Endocarditis patients undergoing valve surgery will also be compared to patients undergoing similar surgery for non-infectious reasons (control group).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-08-06 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic complications | up to 1 year
  Any thromboembolic complications occuring between surgery and 1 year post operatively (incidence, class and severity)

SECONDARY OUTCOMES:
Incidence of perioperative coagulation abnormalities | First 24 hours after surgery
  How often perioperative coagulation abnormalities, measured by classical laboratory values and rotational thromboelastometry are seen from diagnosis to 24 hours post-surgery
Differences in incidence of pathogens and the relation with disease severity | Up to 30 days
  To evaluate the effect of different pathogens (evaluated by laboratory results) on the clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, MD,PhD,PhD, Principal Investigator — Amsterdam Academic Medical Center
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murdoch DR, Corey GR, Hoen B, Miro JM, Fowler VG Jr, Bayer AS, Karchmer AW, Olaison L, Pappas PA, Moreillon P, Chambers ST, Chu VH, Falco V, Holland DJ, Jones P, Klein JL, Raymond NJ, Read KM, Tripodi MF, Utili R, Wang A, Woods CW, Cabell CH; International Collaboration on Endocarditis-Prospective Cohort Study (ICE-PCS) Investigators. Clinical presentation, etiology, and outcome of infective endocarditis in the 21st century: the International Collaboration on Endocarditis-Prospective Cohort Study. Arch Intern Med. 2009 Mar 9;169(5):463-73. doi: 10.1001/archinternmed.2008.603. PMID 19273776
- [Background] Pant S, Patel NJ, Deshmukh A, Golwala H, Patel N, Badheka A, Hirsch GA, Mehta JL. Trends in infective endocarditis incidence, microbiology, and valve replacement in the United States from 2000 to 2011. J Am Coll Cardiol. 2015 May 19;65(19):2070-6. doi: 10.1016/j.jacc.2015.03.518. PMID 25975469
- [Background] Cahill TJ, Prendergast BD. Infective endocarditis. Lancet. 2016 Feb 27;387(10021):882-93. doi: 10.1016/S0140-6736(15)00067-7. Epub 2015 Sep 1. PMID 26341945
- [Background] Durante-Mangoni E, Molaro R, Iossa D. The role of hemostasis in infective endocarditis. Curr Infect Dis Rep. 2014 Nov;16(11):435. doi: 10.1007/s11908-014-0435-8. PMID 25230604
- [Background] Prendergast BD, Tornos P. Surgery for infective endocarditis: who and when? Circulation. 2010 Mar 9;121(9):1141-52. doi: 10.1161/CIRCULATIONAHA.108.773598. No abstract available. PMID 20212293
- [Background] Buyukasyk NS, Ileri M, Alper A, Senen K, Atak R, Hisar I, Yetkin E, Turhan H, Demirkan D. Increased blood coagulation and platelet activation in patients with infective endocarditis and embolic events. Clin Cardiol. 2004 Mar;27(3):154-8. doi: 10.1002/clc.4960270312. PMID 15049384
- [Background] Na S, Shim JK, Chun DH, Kim DH, Hong SW, Kwak YL. Stabilized infective endocarditis and altered heparin responsiveness during cardiopulmonary bypass. World J Surg. 2009 Sep;33(9):1862-7. doi: 10.1007/s00268-009-0107-2. PMID 19597879
- [Background] Thota R, Ganti AK, Subbiah S. Apparent heparin resistance in a patient with infective endocarditis secondary to elevated factor VIII levels. J Thromb Thrombolysis. 2012 Jul;34(1):132-4. doi: 10.1007/s11239-012-0692-z. PMID 22302637
- [Background] Yu S, Khalpey ZI, Wong RK, Huynh T, Nielsen VG. Complete antithrombin replacement for anticoagulation for cardiopulmonary bypass to repair severe infective mitral valve endocarditis. Blood Coagul Fibrinolysis. 2018 Jan;29(1):123-125. doi: 10.1097/MBC.0000000000000668. PMID 28957943
- [Background] Ileri M, Alper A, Senen K, Durmaz T, Atak R, Hisar I, Yetkin E, Turhan H, Demirkan D. Effect of infective endocarditis on blood coagulation and platelet activation and comparison of patients with to those without embolic events. Am J Cardiol. 2003 Mar 15;91(6):689-92. doi: 10.1016/s0002-9149(02)03405-7. PMID 12633799
- [Background] Salis S, Mazzanti VV, Merli G, Salvi L, Tedesco CC, Veglia F, Sisillo E. Cardiopulmonary bypass duration is an independent predictor of morbidity and mortality after cardiac surgery. J Cardiothorac Vasc Anesth. 2008 Dec;22(6):814-22. doi: 10.1053/j.jvca.2008.08.004. Epub 2008 Oct 22. PMID 18948034
- [Background] Salsano A, Giacobbe DR, Sportelli E, Olivieri GM, Natali R, Prevosto M, Del Bono V, Viscoli C, Santini F. Aortic cross-clamp time and cardiopulmonary bypass time: prognostic implications in patients operated on for infective endocarditis. Interact Cardiovasc Thorac Surg. 2018 Sep 1;27(3):328-335. doi: 10.1093/icvts/ivy085. PMID 29579243
- [Background] Dahn H, Buth K, Legare JF, Mingo H, Kent B, Whynot S, Scheffler M. Endocarditis is not an Independent Predictor of Blood Transfusion in Aortic Valve Replacement Patients With Severe Aortic Regurgitation. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):687-91. doi: 10.1053/j.jvca.2015.10.003. Epub 2015 Oct 9. PMID 26750645
- [Background] Deppe AC, Weber C, Zimmermann J, Kuhn EW, Slottosch I, Liakopoulos OJ, Choi YH, Wahlers T. Point-of-care thromboelastography/thromboelastometry-based coagulation management in cardiac surgery: a meta-analysis of 8332 patients. J Surg Res. 2016 Jun 15;203(2):424-33. doi: 10.1016/j.jss.2016.03.008. Epub 2016 Mar 26. PMID 27363652